CLINICAL TRIAL: NCT02777788
Title: Advanced Non-small Cell Lung Cancer With Chinese Medicine Comprehensive Treatment Plan
Brief Title: Curative Study of Chinese Traditional Medicine to Treat Lung Cancer
Acronym: TCM
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Chest Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ZY3-CCCX-3-3023
Record Dates: First submitted 2016-05-09; First posted 2016-05-19 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-05

CONDITIONS: Cancer
Keywords: Chinese Traditional Medicine
MeSH Terms: conditions — Neoplasms | interventions — jinfukang; Pemetrexed; nedaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chemotherapy (Active Comparator): Eligible subjects will be treated with platinum-doublet 2 cycles chemotherapy:pemetrexed,docetaxel,gemcitabine,paclitaxel or vinorelbine combined with carboplatin、cis-platinum or nedaplatin. Each cycle was 21-days.
  Dosage:pemetrexed i.v.500mg/m2 d1 ; docetaxel i.v.75mg/m2 d1 ; gemcitabine i.v.1250 mg/m2 d1,d8 ; paclitaxel i.v.175mg/m2 d1 ; vinorelbine i.v.25mg/m2 d1,d8; carboplatin i.v.area under curve (AUC) 5 d1 ；cis-platinum i.v.75mg/m2 d1（or divided into 3days）；nedaplatin i.v.80mg/m2 d1.
  Interventions: Drug: pemetrexed,docetaxel,gemcitabine,paclitaxel or vinorelbine combined with carboplatin、cis-platinum or nedaplatin
- TCM combined chemotherapy (Experimental): TCM：JinFuKang plus XingZaoRuanJian, chemotherapy will be the same. JinFuKang po.tid.30ml d6-d21 XingZaoRuanJian po.tid.30ml d6-d21
  Interventions: Drug: JinFuKang; Drug: XingZaoRuanJian

INTERVENTIONS:
Drug: JinFuKang — treated with chemotherapy
  Other Names: JinFuKang oral liquid
  Arms: TCM combined chemotherapy
Drug: XingZaoRuanJian — treated with chemotherapy
  Other Names: RuanHuaTang
  Arms: TCM combined chemotherapy
Drug: pemetrexed,docetaxel,gemcitabine,paclitaxel or vinorelbine combined with carboplatin、cis-platinum or nedaplatin
  Arms: chemotherapy

SUMMARY:
The purpose of this study is to observe the efficacy of chemotherapy combined with Chinese patent drugs for patients with advanced non-small-cell lung cancer, also to evaluate the adverse reaction and the reliability.

DETAILED DESCRIPTION:
Lung cancer is the most common malignant tumor in the world with about 80%-85% non small cell lung cancer.

The investigators perform a multi-center, randomized, controlled, prospective study in patients with advanced NSCLC. Patients are randomized over observational group(Chinese patent drugs plus chemotherapy), and control group (chemotherapy). The investigators will observe 2 cycles and after that regular follow-up will be arranged.

The primary end point is: Objective response rate;

The secondary end points are:

1. progression-free survival(PFS);
2. overall survival(OS);
3. Time to Progression (TTP);
4. quality of life questionnaire（QOL);
5. other end points are: Toxicity, side effects and security of the treatments will be assessed at the same time.

The investigators expect that integrated TCM combined with chemotherapy has a better efficacy on enhancing Objective response rate，prolonging PFS, OS, improving QOL, reducing the adverse reaction of patients than that of chemotherapy.Therefore our study can provide evidences for optimizing and promoting integrated TCM combined with Western Medicine treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically confirmed of stage Ⅲb-Ⅳ NSCLC
2. Ages Eligible for Study: 18-65 years old;
3. Physical status score (ECOG PS) ≤ 2 scores；
4. Estimated life expectancy of at least 6 months；
5. Participants have no major organ dysfunction and chemotherapy contraindications: hemoglobin ≥10g/dL, absolute neutrophil count (ANC) ≥1.5*109/L, platelets ≥80*109/L, Liver and kidney function is normal;
6. Informed consent from the patient.

Exclusion Criteria:

1. Patient with other malignant tumor except NSCLC 5 years previous to study entry.
2. Patients who have received targeted drug treatment；
3. Serious problem of heart, liver or kidney with severe dysfunction;
4. Pregnant or child breast feeding women;
5. Mental or cognitive disorders;
6. Participating in other drug trials;
7. Who are allergic to the study drug.
8. Diabetic patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | From date of randomization until the date of first documented progression or date of death from any cause，up to 2 months
  The progression disease is assessed based on CT every 2 months from date of randomization and the endpoints is the date of first documented progression or date of death due to lung cancer.

SECONDARY OUTCOMES:
Objective response rate | up to 2 months
Time-to-Progression | up to 2 months
Number of participants with treatment-related quality of life as assessed by FACT-L4.0 | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: HEGEN LI, Study Director — Shanghai University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: Undecided